CLINICAL TRIAL: NCT06530511
Title: A Prospective, Single-arm, Multicenter Clinical Study of Polatuzumab, Rituximab and Orelabrutinib Combination Regimen (PRO) in the Treatment of Elderly Patients with Frail Treatment-naive Non-germinal Center Subtype Diffuse Large B-cell Lymphoma
Brief Title: Polatuzumab, Rituximab and Orelabrutinib Combination Regimen (PRO) in the Treatment of Elderly Frail Patients with Treatment-naive Non-GCB DLBCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Principal Investigator, Wenyu Shi, Director, Department of Oncology, Affiliated Hospital of Nantong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JCLG-24-7
Record Dates: First submitted 2024-07-23; First posted 2024-07-31 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-07

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: elderly; frail; PRO; Non-GCB; DLBCL
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — polatuzumab vedotin; Rituximab; orelabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PRO (Experimental): The drugs involved in this trial include Polatuzumab, Rituximab, and orelabrutinib in 21-day cycles.
  The dose and administration method of the study drug were as follows:
  * Polatuzumab: 1.8 mg/kg, IV, D1;
  * Rituximab: 375 mg/m2, IV, D1;
  * Orelabrutinib: 150 mg/time, qd, po, D1-21;
  Interventions: Drug: Polatuzumab vedotin; Drug: Rituximab; Drug: Orelabrutinib

INTERVENTIONS:
Drug: Polatuzumab vedotin — Polatuzumab: 1.8 mg/kg, IV Drip infusion, D1;
Drug: Rituximab — Rituximab: 375 mg/m2, IV Drip infusion, D1
Drug: Orelabrutinib — Orelabrutinib: 150 mg/time, qd, po, D1-21

SUMMARY:
This prospective, single-arm, multicenter clinical study aims to enroll 30 frail elderly patients with Non-GCB DLBCL. This study is to evaluate the preliminary efficacy and safety of the combination of Polatuzumab, Rituximab, and orelabrutinib in this population. The primary endpoint is CR rate after induction therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histopathologically confirmed DLBCL;

  * The sGA evaluation result of octogenarians or 60-79 years old is unfit or f RA il;

    * Non-germinal center (Non-GCB) type;

      * ECOG performance status score of 0-3 points; ⑤ No previous treatment for Lymphoma (unless glucocorticoid); 6 Radiographic Investigation to measurable disease, defined as the longest diameter with at least one Lymph node disorder > 1.5 cm, or at least one extranodal lesion > 1.0 cm in the longest diameter; ⑦ Adequate organ function;

        * Life expectancy ≥ 12 weeks; ⑨ Signed written informed consent.

Exclusion Criteria:

* Accompanied by uncontrolled cardiovascular and cerebrovascular diseases, Coagulopathy diseases, autoimmune diseases and severe Immunization diseases, etc.;

  * Laboratory abnormalities at screening (unless caused by Lymphoma) A) ANC < 1.5 x 109/L, PLT < 80 x 109/L b） Coagulation: INR greater than 1.5 x upper limit of normal; PT and APTT greater than 1.5 x upper limit of normal c） Liver function: ALT or AST 2 times higher than upper limit of normal, AKP and Bilirubin 1.5 times higher than upper limit of normal d） Renal function: Creatinine high 1.5 times the upper limit of normal, Creatinine clearance < 60 mL/min (estimated by C OC kcroft-Gault formula); ③ HIV Infection;

    * HbsAg positive patients should be HBV DNA negative before enrollment; in addition, if the patients are HBsAg negative but HBcAb positive (regardless of HBsAb status), HBV DNA detection is still required; if the results are positive, antiviral therapy is required, and HBV DNA negative before enrollment;

      * Requires continuous treatment with strong and moderate CYP3A inhibitors or CYP3A Induction agents. Patients who have taken strong and moderate CYP3A inhibitors or CYP3A Induction agents (or have taken these agents within 5 half-lives) within 7 days prior to the first dose of study drug should not be enrolled; ⑥ Inability to swallow capsules or suffering from diseases that seriously affect gastrointestinal function, such as Syndrome malabsorption, gastric or Small intestinal resection, symptomatic Inflammatory bowel disease or partial or complete Intestinal obstruction; ⑦ Other concurrent and uncontrolled medical conditions that, in the opinion of the investigators, would affect the patients' participation in the study, including patients with Psychosis or other patients known or suspected to be unable to fully comply with the study protocol.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
CRR | 6 months
  Complete response rate (CRR) at the end of Induction treatment (6 cycles)

SECONDARY OUTCOMES:
ORR | 6 months
  Overall response rate (ORR) at the end of Induction treatment (6 cycles)
2y-PFS rate | 24 months
  defined as the time from the start of treatment to the first documented Disease progression or Death; patients who have not experienced an event at the time of analysis will be censored at the date of the most recent disease assessment
OS | 24 months
  defined as the time from the start of treatment to the Death of death from any cause; patients who had not experienced an event at the time of analysis were censored at the date the patient was last known to be alive
EFS | 24 months
  defined as the time from the start of treatment until Disease progression/relapse, Death from any cause, or the start of next-line Lymphoma therapy (NALT); patients who have not experienced an event at the time of analysis will be censored at the date of the most recent disease assessment
Safety profile | 24 months
  defined as the incidence of Adverse event (AEs) that occurred from the date of the first dose of Carcinoma until 30 days after discontinuation of study drug or PD or initiation of new anti-safety therapy, whichever occurred first, and defined as all Adverse event that occurred after the patient received the study regimen; defined as the incidence of treatment-related AEs that were considered by the investigator to be related to Salvage therapy, Transplant, and consolidation therapy after the patient received the study regimen

OTHER OUTCOMES:
Potential predictive factors | 24 months
  defined as clinical and biological factors at baseline or during the treatment that might be associated with treatment efficacy and safety and was performed to screen out populations that would benefit more from this protocol.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Affiliated hospital of Nantong University, Nantong, Jiangsu
  - Jiangsu Province Hospital, Nanjing

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting 6 months after publication
Access Criteria: IPD could be shared by contacting the corresponding author via email after publication